CLINICAL TRIAL: NCT07087548
Title: Chronic Lumbar Disc Herniation: A Randomized Single-Blind Study on the Comparative Efficacy of Peloid Therapy Versus Hot Pack Therapy
Brief Title: A Study Comparing Peloid Therapy and Hot Pack Treatment in Adults With Chronic Low Back Pain Caused by Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, assistant professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/324
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2021-09

CONDITIONS: Lumbal Disc Herniation
MeSH Terms: interventions — Mud Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Peloid Therapy+TENS) (Experimental): The peloid therapy group received 15 sessions of peloid therapy at 45°C for 30 minutes per session, five days a week for three weeks. Peloid was applied to the lumbar region with a brush to a thickness of approximately 15 mm. The area was then wrapped with stretch film and a towel for 30 minutes to minimize heat loss. Peloids produced and packaged in the Afyonkarahisar Sandıklı geothermal region were used. The peloid is gray, odorless, and has a pH of 8.74. It contains humic acid, humin, lignin, hemicellulose, montmorillonite, calcite, and kaolinite. After the peloid application, the area was cleaned, and conventional TENS (80 Hz frequency) was applied to the waist for 20 minutes.
  Interventions: Other: Peloid Therapy
- Hot pack Therapy (Hotpack+TENS) (Active Comparator): The hot pack group applied 20 minutes, 5 days a week, once a day, for 15 sessions on the lumbar region. The boiler temperature of the hot packs used was 90 °C. Two towels were used, with the thickest side of the towels placed on the lumbar area of the individuals. Then, conventional TENS (80 Hz frequency) was applied to the painful area in the lumbar region for 20 minutes
  Interventions: Other: Hotpack Therapy

INTERVENTIONS:
Other: Peloid Therapy — Peloid therapy will be applied using medical mud packs at 45°C for 30 minutes per session, 5 sessions per week for 3 consecutive weeks. The therapy will be administered to the lower back region in patients diagnosed with chronic lumbar disc herniation. This intervention aims to reduce pain and improve function through thermomechanical and biochemical effects of natural peloid.
  Arms: Experimental (Peloid Therapy+TENS)
Other: Hotpack Therapy — The hot pack group applied 20 minutes, 5 days a week, once a day, for 15 sessions on the lumbar region. The boiler temperature of the hot packs used was 90 °C. Two towels were used, with the thickest side of the towels placed on the lumbar area of the individuals. Then, conventional TENS (80 Hz frequency) was applied to the painful area in the lumbar region for 20 minutes
  Arms: Hot pack Therapy (Hotpack+TENS)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of peloid therapy versus hot pack therapy in adults aged 18-50 with chronic lumbar disc herniation (LDH). The main questions it aims to answer are:

Does peloid therapy reduce pain more effectively than hot pack therapy in patients with chronic LDH?

Does peloid therapy improve functional status, range of motion, and quality of life more than hot pack therapy? Researchers will compare peloid therapy (45°C for 30 minutes, 5 days/week) to hot pack therapy (20 minutes, 5 days/week) to see which treatment offers better clinical outcomes.

Participants will:

Receive either peloid therapy or hot pack therapy for 3 weeks (15 sessions total).

Undergo standard TENS therapy (20 minutes to the lumbar region) after each session.

Complete assessments before and after treatment including:

Pain intensity (Visual Analog Scale - VAS) Functional status (Back Pain Functional Scale - BPFS) Disability level (Oswestry Disability Index - ODI) Quality of life (Short Form-36 - SF-36) Lumbar range of motion and finger-to-floor distance (FFD)

DETAILED DESCRIPTION:
Chronic lumbar disc herniation (LDH) is a common spinal disorder that causes pain, functional limitations, and reduced quality of life. Non-invasive physical therapy modalities such as thermotherapy and electrotherapy are frequently used in conservative management. Peloid therapy, a form of thermal mud treatment, has been proposed to exert anti-inflammatory, analgesic, and muscle-relaxing effects. However, limited controlled studies have compared its clinical effectiveness with more commonly used superficial heat modalities like hot packs.

This single-blind, randomized controlled trial was designed to evaluate and compare the effects of peloid therapy and hot pack therapy in adults diagnosed with chronic LDH. A total of 60 participants were randomly allocated into two treatment arms. The peloid group received a localized application of therapeutic mud (peloid) at 45°C for 30 minutes per session, five days per week for three weeks (total 15 sessions). The control group received conventional hot pack therapy for 20 minutes under the same session frequency and duration. Both groups additionally received transcutaneous electrical nerve stimulation (TENS) to the lumbar region following each thermotherapy session.

Outcome measures were recorded before and after the intervention period and included pain intensity (VAS), functional ability (BPFS), disability index (ODI), quality of life (SF-36), lumbar range of motion (flexion, extension, lateral flexion, and rotation), and finger-to-floor distance (FFD). Statistical analysis was performed to assess within-group and between-group changes.

This study provides comparative data on the efficacy of peloid therapy and conventional hot pack application in a homogeneous patient population with chronic LDH and may inform future guidelines on the selection of conservative treatment modalities in physical therapy practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18 years old with CLBP due to LDH lasting more than three months
* Individuals who showed degeneration and prolapsed herniation on magnetic resonance imaging
* Individuals were examined by a specialist physician

Exclusion Criteria:

* having not received physiotherapy for LDH in the last 6 months,
* severe neurological deficit,
* osteoporosis,
* malignancy, inflammatory disease
* decompensated cardiopulmonary disease,
* uncontrolled hypertension,
* those with an important pathology in routine laboratory tests (liver and kidney dysfunction, individuals with thyroid dysfunction, diabetes),
* vertebral fracture,
* lumbar listhesis
* infectious disease at lumbar level,
* inflammatory lumbar pain,
* individuals with extruded and sequestered herniation as a result of MRI,
* those with neurological deficits,
* communication problems,
* being allergic to peloid or hotpack
* pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Pain intensity (VAS) | Before treatment and after treatment (3rd week).
  Pain severity was assessed with the Visual Analog Scale (VAS), which is scored between 0 and 10, and is used to evaluate pain. 0 denotes no pain and 10 denotes unbearably severe pain. Participants were instructed to indicate the level of pain they experienced by marking a point along a 10 cm straight line, and the value found was recorded in cm

SECONDARY OUTCOMES:
Impact of daily activities on a person's life (Oswestry Disability Index) | before treatment and after treatment (3rd week)
  The Oswestry Disability Index (ODI) is an evaluation questionnaire that assesses the impact of daily activities on a person's life. It has 10 subgroups, each with 6 questions scored from 0 to 5. The subgroups cover pain severity, self-care, lifting-carrying, walking, sitting, standing, sleep, sexual life, travel, and social life. The total score ranges from 0 to 50, with higher scores indicating a greater disability.
Assessing functional loss due to low back pain (Back Pain Functional Scale ) | before treatment and after treatment (3rd week)
  The Back Pain Functional Scale (BPFS), is an easy-to-use tool developed by WHO for assessing functional loss due to low back pain, completed by the participant. It evaluates the impact on work, school, home activities, habits, bending, wearing shoes or socks, lifting, sleeping, sitting, standing, walking, climbing stairs, and driving (or traveling if the participant does not drive). Each item is scored from 0 to 5, with 0 indicating the activity is impossible and 5 indicating no difficulty. The total score ranges from 0 to 60, with 60 indicating no difficulty in any activity.
Quality of Life (SF-36) | before treatment and after treatment (3rd week)
  The Short Form Health Survey (SF-36), is a scale consisting of 36 items and measures eight health dimensions: physical function, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty, and mental health. It evaluates the last four weeks, with higher SF-36 scores indicating a better health-related quality of life. Scores range from 0 (worst health) to 100 (best health)
Active ROM measurements (flexion, extension, left and right lateral flexion, and rotation) | before treatment and after treatment (3rd week)
  Active ROM measurements (flexion, extension, left and right lateral flexion, and rotation) of individuals were done with a universal goniometer. Kendall and Mccreary's system was based on the value of degrees. Measurements were taken with participants standing, repeated three times without causing fatigue.
Finger-floor distance measurement | before treatment and after treatment (3rd week)
  Finger-floor distance (FFD) measurement is used for trunk flexibility and mobility. Currently, there is no unified reference value range for FFD measurement. Values of 0 or close to 0 typically indicate good spinal mobility, while higher values usually suggest abnormal or pathological spinal mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Sancak Tıp Merkezi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT07087548/Prot_SAP_000.pdf